CLINICAL TRIAL: NCT01387399
Title: Phase I Study of Intraoperative Hyperthermic Intraperitoneal Chemoperfusion With Cisplatin in Patients With Recurrent Ovarian Cancer
Brief Title: Safety and Pharmacokinetics of Intraoperative Hyperthermic Intraperitoneal Chemoperfusion (HIPEC) With Cisplatin to Treat Platinum-sensitive Recurrent Ovarian Cancer
Acronym: HIPEC ROC I
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Oliver Zivanovic, Priv. Doz. Dr. med. Oliver Zivanovic, University Hospital, Bonn
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT No.: 2010-024652-28
Record Dates: First submitted 2011-06-24; First posted 2011-07-04 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; recurrence; platinum-sensitive recurrent ovarian cancer; HIPEC; intraperitoneal chemotherapy; hyperthermic intraperitoneal chemoperfusion; cisplatin
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin as HIPEC (Experimental): Phase I dose escalating study of cisplatin administered intraoperatively as hyperthermic intraperitoneal chemoperfusion
  Interventions: Procedure: Cisplatin administered intraoperatively as hyperthermic intraperitoneal chemoperfusion

INTERVENTIONS:
Procedure: Cisplatin administered intraoperatively as hyperthermic intraperitoneal chemoperfusion — Classical "3+3" dose escalation study of cisplatin administered as HIPEC (60mg/m², 80mg/m² and 100mg/m²)

SUMMARY:
The purpose of this phase I study is to determine the safety, feasibility, maximum tolerated dose (MTD), pharmacokinetics and pharmacodynamics of Cisplatin administered as Intraoperative Hyperthermic Intraperitoneal Chemoperfusion (HIPEC) in Patients with Platinum-Sensitive Recurrent Ovarian Cancer.

DETAILED DESCRIPTION:
This is a phase I dose escalating study designed to identify tolerable, clinically active doses of cisplatin delivered as intraoperative intraperitoneal hyperthermic chemoperfusion (HIPEC) in patients with platinum-sensitive recurrent ovarian cancer. After surgical cytoreduction, a single dose of cisplatin will be administered in 3 liters normal saline via intraperitoneal HIPEC with closed-abdomen technique for 90 minutes in the hyperthermic phase (41-43 degrees C). After completion of perfusion, the perfusate will be drained, the abdomen opened and the abdomen and pelvis irrigated with 2-3 liters normal saline to wash away any residual chemotherapeutic agent. Fascia and skin will then be closed in a standard fashion. Cisplatin infusion will be discontinued for unacceptable toxicity. The primary objective is to determine the maximum tolerated dose (MTD) of cisplatin administered as HIPEC. Secondary objectives are to determine pharmacokinetics and pharmacodynamics as well as the effect of cisplatin as HIPEC on the ability to subsequently administer 6 cycles of standard platinum-based systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* only female participants are being studied
* signed informed consent
* patients with histologically proven or suspicious recurrent epithelial ovarian cancer (based on Response Evaluation Criteria in Solid Tumors (RECIST)- or CA-125 criteria)
* Progression-free interval after completion of adjuvant platinum-based chemotherapy of 6 months or more.
* Subjects with the following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, adenocarcinoma N.O.S.
* Patients are eligible if the disease is deemed operable to equal or less than 1 cm at the completion of surgery.

Exclusion Criteria:

* mucinous Ovarian cancer
* non-invasive Borderline tumor
* subjects who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin are permitted, provided that it was completed more than 3 years prior to enrollment, and the subject remains free of recurrent or metastatic disease
* subjects with active infection that requires parenteral antibiotics
* patients with any underlying cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions, chronic or latent infectious diseases, immune deficiency, or history, which in the opinion of the investigator, places the patient at an unacceptable risk for participation in the study
* patients with known platinum allergy
* evidence of extensive intraperitoneal adhesions at the time of surgery, as determined by the operating surgeon

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | within the first 21days after surgery
  To determine the safety and maximum tolerated dose (MTD) of cisplatin (60 mg/m², 80mg/m² and 100 mg/m²) administered as intraperitoneal hyperthermic chemoperfusion defined by the dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Pharmacokinetics | within 24 hours of HIPEC
  Blood and peritoneal concentrations of cisplatin will be measured at various time points within the first 24 hours after HIPEC. The elimination half-life and the area under the plasma concentration time curve of cisplatin will be measured. Peritoneal and systemic clearance and distribution of cisplatin will be modeled in a compartmental model.
Number of cycles of standard intravenous platinum-based systemic chemotherapy | 3 months
  Measure the effect of cisplatin as HIPEC on the ability to subsequently administer 6 cycles of standard intravenous platinum-based systemic chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Zivanovic, MD, Principal Investigator — University Hospital, Bonn
Locations (1):
- University Hospital, Bonn, Germany